CLINICAL TRIAL: NCT03054688
Title: Somnotouch-NIBP Compared to Standard Ambulatory 24 Hours Blood Pressure Measurement
Acronym: VAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03061989
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Somnotouch NIBP (Experimental): Blood pressure measurement with Somnotouch-NIBP device in addition to standard cuff based device
  Interventions: Device: Somnotouch NIBP

INTERVENTIONS:
Device: Somnotouch NIBP — Somnotouch NIBP in addition to standard blood pressure measurement

SUMMARY:
Comparison of 24 hours blood pressure measurement with puls-transit time versus cuffs.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent

Exclusion Criteria:

* Atrial fibrillation
* Medical reasons why blood pressure measurement is not possible at the upper extremity (Shunt, Lymphedema)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Difference in mean 24h systolic blood pressure | 24 hours
  Difference in mean 24h systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Burkard, MD, Principal Investigator — University Hospital, Basel, Switzerland; Philipp Krisai, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derendinger FC, Vischer AS, Krisai P, Socrates T, Schumacher C, Mayr M, Burkard T. Ability of a 24-h ambulatory cuffless blood pressure monitoring device to track blood pressure changes in clinical practice. J Hypertens. 2024 Apr 1;42(4):662-671. doi: 10.1097/HJH.0000000000003667. Epub 2024 Jan 23. PMID 38288945
- [Derived] Krisai P, Vischer AS, Kilian L, Meienberg A, Mayr M, Burkard T. Accuracy of 24-hour ambulatory blood pressure monitoring by a novel cuffless device in clinical practice. Heart. 2019 Mar;105(5):399-405. doi: 10.1136/heartjnl-2018-313592. Epub 2018 Sep 18. PMID 30228251